CLINICAL TRIAL: NCT02730351
Title: 201832: A Randomised, Double-Blind, Double-Dummy, Crossover Comparison of Fluticasone Furoate/Vilanterol 100/25 mcg Once Daily Versus Fluticasone Propionate 250 mcg Twice Daily in Adolescent and Adult Subjects With Asthma and Exercise-Induced Bronchoconstriction
Brief Title: Crossover Study Comparing Fluticasone Furoate (FF)/Vilanterol (VI) Once Daily Versus Fluticasone Propionate (FP) Twice Daily in Subjects With Asthma and Exercise-Induced Bronchoconstriction (EIB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201832; 2017-001516-11 (EudraCT Number)
Record Dates: First submitted 2016-03-24; First posted 2016-04-06 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Fluticasone furoate; activity monitoring; Vilanterol; Cross-over; exercise-induced bronchoconstriction; exercise challenge; double-dummy; asthma; spirometry; fluticasone propionate
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/VI 100/25 mcg + Placebo DISKUS®/ ACCUHALER® (Experimental): Randomised subjects will receive FF/VI 100/25 mcg once daily via ELLIPTA inhaler and placebo twice daily via DISKUS / ACCUHALER for 2 weeks in Period 1. There will be a washout period of 2 weeks between treatment periods in which subjects will receive FP 250 mcg twice daily. Subjects will receive FP 250 mcg twice daily via DISKUS inhaler and placebo once daily via ELLIPTA inhaler for 2 weeks in Period 2.
  Interventions: Drug: Fluticasone furoate/ Vilanterol 100 mcg/25 mcg; Drug: Placebo via DISKUS / ACCUHALER
- FP 250 mcg + Placebo ELLIPTA® (Experimental): Randomised subjects will receive FP 250 mcg twice daily via DISKUS inhaler and placebo once daily via ELLIPTA inhaler for 2 weeks in Period 1. There will be a washout period of 2 weeks between treatment periods in which subjects will receive FP 250 mcg twice daily. Subjects will receive FF/VI 100/25 mcg once daily via ELLIPTA inhaler and placebo twice daily via DISKUS inhaler for 2 weeks in Period 2.
  Interventions: Drug: Fluticasone propionate 250 mcg; Drug: Placebo via ELLIPTA inhaler

INTERVENTIONS:
Drug: Fluticasone furoate/ Vilanterol 100 mcg/25 mcg — FF/VI 100/25 mcg will be administered via ELLIPTA inhaler once daily in the evening
  Arms: FF/VI 100/25 mcg + Placebo DISKUS®/ ACCUHALER®
Drug: Fluticasone propionate 250 mcg — FP 250mcg will be administered via DISKUS inhaler, twice daily, once in the morning and once in the evening
  Arms: FP 250 mcg + Placebo ELLIPTA®
Drug: Placebo via ELLIPTA inhaler — Placebo will be administered via ELLIPTA inhaler once daily in the evening
  Arms: FP 250 mcg + Placebo ELLIPTA®
Drug: Placebo via DISKUS / ACCUHALER — Placebo will be administered via DISKUS / ACCUHALER, twice daily, once in the morning and once in the evening
  Arms: FF/VI 100/25 mcg + Placebo DISKUS®/ ACCUHALER®

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, crossover study with two 2-week treatment periods separated by a 2-week wash-out period. Subjects will participate in up to eight study visits and have a follow up phone call approximately a week after the last clinic visit. Visits 1, 2, 3, 5 and 6 are evening visits that will be conducted between 5PM and 11PM. Visit 4 and Visit 7 are also evening visits that will begin between 5PM and 11PM and continue over a period of approximately 24 hours. Subjects will be required to attend three clinic visits during this 24-hour period. An exercise challenge (using a treadmill) will be conducted at Visit 2, Visit 3 and Visit 6 (after 23 hours of the first treatment dose in each Treatment Period); and at 12 and 23 hours post evening dose at Visits 4 and 7. Spirometry will be conducted at specified visits and prior to and after each exercise challenge.

Subjects with symptomatic allergic rhinitis at Visit 1 (screening) may be treated for up to four weeks with intranasal corticosteroids followed by a repeat screening visit to determine eligibility prior to entry into the study.

Eligible subjects at visit 1 will complete a 4-week single blind run-in on FP 250 microgram (mcg) twice daily (BID), followed by 2-week double-blind Treatment Period 1 on randomized treatment, a 2-week single blind washout period on FP 250 mcg BID, 2-week double-blind Treatment Period 2 receiving the alternative treatment, and follow-up contact approximately 7-days after completing Treatment Period 2. The total duration of study participation is approximately 11 weeks; and up to 15 weeks for subjects with Symptomatic Allergic Rhinitis.

The primary objective of the study is to evaluate the protective effect of fluticasone furoate/vilanterol (FF/VI) 100/25 mcg once-daily compared with fluticasone propionate (FP) 250 mcg twice-daily against exercise-induced bronchoconstriction in adolescent and adult subjects aged 12 to 50 with persistent asthma.

ELLIPTA, ACCUHALER, and DISKUS are registered trademarks of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Subjects must give their signed and dated written informed consent to participate prior to commencing any study related activities.
* Age Range: 12 to 50 years of age, inclusive, at Visit 1 (Screening).
* Diagnosis: A diagnosis of asthma, as defined by the National Institutes of Health for at least 12 weeks prior to Visit 1.
* Asthma Severity: Subjects must have a pre-bronchodilator FEV1 of >=70 percent of the predicted normal value. Predicted values will be based upon Global Lung Function Initiative equations for spirometry reference values.
* Evidence of EIB: Subjects must answer "Yes" to at least 2 of the following 3 questions reflecting on the previous 12 months:

  * Are you short of breath during exercise or other physical exertion?
  * Do you wheeze after exercise or other physical exertion?
  * Do you cough after exercise or other physical exertion?
* Concurrent Anti-Asthma Therapy: Subjects must be taking low- to moderate dose inhaled steroids for 12 weeks prior to Visit 1 in order to participate with no change in dose for the 4 weeks prior to Visit 1.
* Gender: Subjects may be male or an eligible female. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile).Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, > 45 years, in the absence of hormone replacement therapy.

OR Child bearing potential, has a negative pregnancy test at screening, and agrees to acceptable contraceptive methods approved in their local country, when used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact).

* Albuterol/salbutamol Use: All subjects must be able to replace their current short-acting beta2-agonist with albuterol/salbutamol, to be used only on an as-needed basis for the duration of the study. Each subject must be judged capable of withholding albuterol/salbutamol for at least 6 hours prior to performing spirometric evaluations.
* Physical Capacity: Each subject must be physically able to perform the exercise challenges on a treadmill when bronchodilators have been withheld.

Exclusion Criteria:

* Intermittent Asthma, Seasonal Asthma, or Exercise-Induced Bronchoconstriction Only: Subjects with only intermittent or seasonal asthma or only exercise-induced asthma are excluded from participation in this study.
* History of Life-threatening Asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 10 years.
* Asthma Exacerbation: Any asthma exacerbation requiring oral corticosteroids within 12 weeks of Visit 1 or that resulted in an overnight hospitalization requiring additional treatment for asthma within 6 months prior to Visit 1.
* Symptomatic Allergic Rhinitis: Subjects with symptomatic allergic rhinitis at Visit 1 may be treated for up to four weeks with intranasal corticosteroids followed by a repeat screening visit to determine eligibility prior to entry into the study. Subjects that continue to be symptomatic after up to four weeks of treatment will be excluded.
* 12-Lead Electrocardiogram (ECG): A subject is not eligible if he/she has an abnormal, clinically significant ECG as determined by the investigator at the Screening Visit.
* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 and led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Concurrent Respiratory Disease: A subject must not have current evidence of:

  1. Atelectasis 2. Bronchopulmonary dysplasia 3. Chronic bronchitis 4. Chronic obstructive pulmonary disease (COPD) (current or past diagnosis including asthma/COPD overlap) 5. Pneumonia 6. Pneumothorax 7. Interstitial lung disease 8. Or any evidence of concurrent respiratory disease other than asthma.
* Other Concurrent Diseases/Abnormalities: A subject must not have any clinically significant, uncontrolled condition, or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
* Investigational Medications: A subject must not have used any investigational drug within 30 days prior to Visit 1 or within five half-lives (t1/2) of the prior investigational study, whichever is longer of the two periods.
* Allergies: 1) Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy, or excipients used with FF/VI 100/25 or FP 250 (i.e., drug, lactose or magnesium stearate). 2) Milk Protein Allergy: History of severe milk protein allergy. 3) Latex Allergy: History of allergy or sensitivity to latex that in the opinion of the investigator contraindicates the subject's participation in the study.
* Concomitant Medication: Administration of prescription or non-prescription medication that would significantly affect the course of asthma, or interact with study drug.
* Immunosuppressive Medications: A subject must not be using or require the use of immunosuppressive medications during the study.
* Compliance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, disease, or geographical location which seems likely (in the opinion of the investigator) to impair compliance with any aspect of this study protocol.
* Tobacco/Marijuana Use: Current tobacco smoker or has a smoking history of >=10 pack-years (20 cigarettes/day for 10 years). A subject may not have used inhaled tobacco products or inhaled marijuana within the past 3 months (e.g. cigarettes, cigars, electronic cigarettes, or pipe tobacco).
* Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study-coordinator or an employee of the participating investigator.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (12):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, El Paso, Texas
- Canada (2):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Mississauga, Ontario

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=201832

REFERENCES:
- [Background] Martin N, Weiler JM, Pearlman D, Jacques L, Nunn C, Forth R, West S, Dunn K, O'Byrne PM. Fluticasone furoate/vilanterol versus fluticasone propionate in patients with asthma and exercise-induced bronchoconstriction. J Asthma. 2020 Apr;57(4):431-440. doi: 10.1080/02770903.2019.1579344. Epub 2019 Feb 22. PMID 30795705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, double-dummy, crossover comparison study of fluticasone furoate (FF)/vilanterol (VI) versus fluticasone propionate (FP) in adolescent and adult participants with asthma and exercise-induced bronchoconstriction (EIB). The study was conducted in two countries-United States and Canada.
Pre-assignment Details: The study consisted of 4-week single-blind run-in, 2-week double-blind treatment period 1, 2-week single-blind wash out, 2-week double-blind treatment period 2 and 1-week Follow-up. A total of 163 participants were screened, 75 were randomized and 74 were included in Intent-To-Treat (ITT) Population who received at least 1 dose of trial medication.
Groups:
- FF/VI 100/25 µg Followed by FP 250 µg: After screening, the eligible participants entered a 4-week single blind run-in period on FP 250 microgram (µg) twice daily (BID) following which the participants were randomized to receive FF/VI 100/25 µg once daily (QD) via ELLIPTA + Placebo BID via DISKUS in treatment period 1 followed by a 2-week single blind wash-out period on FP 250 µg BID. The participants then received FP 250 µg BID via DISKUS + Placebo QD via ELLIPTA in treatment period 2. The participants were followed up for approximately 7 days after completing Treatment Period 2. Albuterol/salbutamol was issued for rescue use during the run-in, wash-out and treatment periods as needed.
- FP 250 µg Followed by FF/VI 100/25 µg: After screening, the eligible participants entered a 4-week single blind run-in period on FP 250 µg BID following which the participants were randomized to receive FP 250 µg BID via DISKUS + Placebo QD via ELLIPTA in treatment period 1 followed by a 2-week single blind wash-out period on FP 250 µg BID. The participants then received FF/VI 100/25 µg QD via ELLIPTA + Placebo BID via DISKUS in treatment period 2. The participants were followed up for approximately 7 days after completing Treatment Period 2. Albuterol/salbutamol was issued for rescue use during the run-in, wash-out and treatment periods as needed.
Period: Treatment Period 1 (2 Weeks)
Arm/Group | FF/VI 100/25 µg Followed by FP 250 µg | FP 250 µg Followed by FF/VI 100/25 µg
Started | 37 | 37
Completed | 36 | 37
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Wash-out Period (2 Weeks)
Arm/Group | FF/VI 100/25 µg Followed by FP 250 µg | FP 250 µg Followed by FF/VI 100/25 µg
Started | 36 | 37
Completed | 35 | 36
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment Period 2 (2 Weeks)
Arm/Group | FF/VI 100/25 µg Followed by FP 250 µg | FP 250 µg Followed by FF/VI 100/25 µg
Started | 35 | 36
Completed | 33 | 36
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treatment Combined: After screening, the eligible participants entered a 4-week single blind run-in period on FP 250 µg BID following which the participants were randomized to one of the following two treatment sequences in a ratio of 1:1: FF/VI 100/25 µg QD via ELLIPTA + Placebo BID via DISKUS in treatment period 1 followed by FP 250 µg BID via DISKUS + Placebo QD via ELLIPTA in treatment period 2 or FP 250 µg BID via DISKUS + Placebo QD via ELLIPTA in treatment period 1 followed by FF/VI 100/25 µg once daily (QD) via ELLIPTA + Placebo BID via DISKUS in treatment period 2. All participants entered a 2-week single blind wash-out period on FP 250 µg BID between the two treatment periods. The participants were followed up for approximately 7 days after completing Treatment Period 2. Albuterol/salbutamol was issued for rescue use during the run-in, wash-out and treatment periods as needed.
Arm/Group | All Treatment Combined
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: African American/African Heritage | 28
  Race, Customized: Asian - South East Asian Heritage | 3
  Race, Customized: White - White/Caucasian/European Heritage | 42
  Race, Customized: Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximal Percent Decrease in Forced Expiratory Volume in One Second (FEV1) Following Exercise Challenge at 12 Hours (Hrs) Post Evening Dose From Pre-exercise FEV1.
Description: The exercise challenge test is a stepped challenge on a treadmill. It was performed at 12 hrs post evening dose at the end of the 2-week treatment period, wherein the participants exercised sufficiently to reach a heart rate between 80 to 95 percent of their predicted maximum within 4 minutes (min) and maintained the heart rate with exercise for an additional 6 min followed immediately by serial assessments of FEV1 at 5, 10, 15, 30, 45 and 60 min post-exercise. Maximal percent decrease was calculated as pre-exercise FEV1 minus minimum post exercise FEV1 (smallest FEV1 value collected within one hr following exercise challenge) divided by pre-exercise FEV1 multiplied by 100. Pre-exercise FEV1 was defined as the FEV1 collected prior to the exercise challenge test at 12 hr post dose. ITT Population comprised of all participants randomized to treatment and who received at least one dose of study medication.
Time Frame: At Week 2 of treatment period 1 and 2
Population: ITT Population. Participants with non-missing covariates and data specific to endpoint were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percentage of FEV1
Groups:
- FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS: Participants were administered FF/VI 100/25 µg QD via ELLIPTA + Placebo BID via DISKUS in one of the two treatment periods. Each treatment period was of 2 weeks with a single blind 2 week wash-out period on FP 250 µg BID between the treatment periods. Albuterol/salbutamol was issued for rescue use during the run-in, wash-out and treatment periods as needed.
- FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA: Participants were administered FP 250 µg BID via DISKUS + Placebo QD via ELLIPTA in one of the two treatment periods. Each treatment period was of 2 weeks with a single blind 2 week wash-out period on FP 250 µg BID between the treatment periods. Albuterol/salbutamol was issued for rescue use during the run-in, wash-out and treatment periods as needed.
Arm/Group | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA
Number analyzed (Participants) | 70 | 69
Percentage of FEV1 | 15.02 (1.058) | 16.71 (1.095)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS vs FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA; Test type: Other; p = 0.109, Mixed Models Analysis — Mixed model repeated measures analysis adjusted for fixed effects of treatment, sex, age, treatment period, smoking history, period Baseline FEV1 and the mean of the two period Baseline FEV1 values. Subject is fitted as a random effect; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-3.76 to 0.39]

2. Secondary Outcome: Maximal Percent Decrease in FEV1 Following Exercise Challenge at 23 Hrs Post Evening Dose From Pre-exercise FEV1.
Description: The exercise challenge test is a stepped challenge on a treadmill. It was performed at 23 hrs post evening dose at the end of the 2-week treatment period, wherein the participants exercised sufficiently to reach a heart rate between 80 to 95 percent of their predicted maximum within 4 min and maintained the heart rate with exercise for an additional 6 min followed immediately by serial assessments of FEV1 at 5, 10, 15, 30, 45 and 60 min post-exercise. Maximal percent decrease was calculated as pre-exercise FEV1 minus minimum post exercise FEV1 (smallest FEV1 value collected within one hr following exercise challenge) divided by pre-exercise FEV1 multiplied by 100. Pre-exercise FEV1 was defined as the FEV1 collected prior to the exercise challenge test at 23 hr post dose.
Time Frame: At Week 2 of treatment period 1 and 2
Population: ITT Population. Participants with non-missing covariates and data specific to endpoint were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percentage of FEV1
Arm/Group | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA
Number analyzed (Participants) | 68 | 69
Percentage of FEV1 | 11.90 (1.020) | 14.05 (1.051)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS vs FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA; Test type: Other; p = 0.051, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-4.31 to 0.01]

3. Secondary Outcome: Proportion of Participants With a 30 Min Post-challenge FEV1 no More Than 5 Percent Lower Than Pre-exercise FEV1 Following the Exercise Challenge at 12 Hrs and 23 Hrs Post Evening Dose.
Description: The blinded treatment exercise challenge test was performed at the end of 2-weeks of treatment period 1 and treatment period 2 on a treadmill at 12 hrs and 23 hrs after administration of the evening dose of study treatment. The challenge was followed immediately by serial assessments of FEV1 at 5, 10, 15, 30, 45 and 60 min post-exercise. Pre-exercise FEV1 was defined as the FEV1 value collected prior to the exercise challenge test at 23 hrs post-dose. Number of participants listed is the number in the ITT population. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: At Week 2 of treatment period 1 and 2
Population: ITT Population. Participants with non-missing covariates and data specific to endpoint were analyzed
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA
Number analyzed (Participants) | 73 | 72
Participants
  FEV1 >=95% of pre-exercise FEV1, 12 hrs; n=70, 69: number analyzed (Participants) | 70 | 69
  FEV1 >=95% of pre-exercise FEV1, 12 hrs; n=70, 69 | 34 | 29
  FEV1 < 95% of pre-exercise FEV1, 12 hrs; n=70, 69: number analyzed (Participants) | 70 | 69
  FEV1 < 95% of pre-exercise FEV1, 12 hrs; n=70, 69 | 36 | 40
  FEV1 >=95% of pre-exercise FEV1, 23 hrs; n=68, 69: number analyzed (Participants) | 68 | 69
  FEV1 >=95% of pre-exercise FEV1, 23 hrs; n=68, 69 | 42 | 37
  FEV1 < 95% of pre-exercise FEV1, 23 hrs; n=68, 69: number analyzed (Participants) | 68 | 69
  FEV1 < 95% of pre-exercise FEV1, 23 hrs; n=68, 69 | 26 | 32
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS vs FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA; Test type: Other; p = 0.266, Regression, Logistic — Repeated measures logistic regression model with parameters estimated using the Generalized Estimating Equation method. Covariates of treatment, sex, age, treatment period, and period baseline FEV1 were included; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.80 to 2.26] — 12 hrs: modeling the odds of having FEV1 >/=95% of pre exercise FEV1 at each of the two time points
Statistical Analysis 2: Comparison: FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS vs FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA; Test type: Other; p = 0.322, Regression, Logistic — Repeated measures logistic regression model with parameters estimated using the Generalized Estimating Equation method; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.73 to 2.58] — 23 hrs: modeling the odds of having FEV1 >/=95% of pre exercise FEV1 at each of the two time points

4. Secondary Outcome: Weighted Mean 0-60 Min for Percentage Decrease From Pre-exercise FEV1 Following Exercise Challenge at 12 Hrs and 23 Hrs Post Evening Dose.
Description: The exercise challenge testing at the end of 2 week treatment period was performed on a treadmill at 12 hrs and 23 hrs after administration of the evening dose of double-blind treatment. Following exercise challenge testing, post-exercise FEV1 values were assessed serially at 5, 10, 15, 30, 45 and 60 min. Pre-exercise FEV1 was defined as the FEV1 value collected prior to the exercise challenge test at 23 hrs post-dose. Number of participants listed is the number in the ITT population. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: At Week 2 of treatment period 1 and 2
Population: ITT Population. Participants with non-missing covariates and data specific to endpoint were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percentage of FEV1
Arm/Group | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA
Number analyzed (Participants) | 73 | 72
Percentage of FEV1
  12 hrs post-dose; n=67, 66: number analyzed (Participants) | 67 | 66
  12 hrs post-dose; n=67, 66 | 5.87 (0.663) | 6.52 (0.680)
  23 hrs post-dose; n=68, 67: number analyzed (Participants) | 68 | 67
  23 hrs post-dose; n=68, 67 | 3.98 (0.699) | 5.73 (0.747)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS vs FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA; Test type: Other; p = 0.342, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-2.01 to 0.71] — 12 hrs post-dose
Statistical Analysis 2: Comparison: FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS vs FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA; Test type: Other; p = 0.041, Mixed Models Analysis — Mixed model repeated measures analysis adjusted for fixed effects of treatment, sex, age, treatment period, smoking history, period Baseline FEV1 and the mean of the two period Baseline FEV1 values; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-3.42 to -0.07] — 23 hrs post-dose

ADVERSE EVENTS:
Time Frame: The on-treatment adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment until the follow-up contact (approximately up to 51 days).
Description: ITT Population
Groups:
- FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS: FF/VI 100/25 µg QD via ELLIPTA + Placebo BID via DISKUS
- FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA: FP 250 µg BID via DISKUS + Placebo QD via ELLIPTA
Arm/Group | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/72
Serious Adverse Events (participants affected / at risk) | 1/73 | 0/72
Other Adverse Events (participants affected / at risk) | 5/73 | 4/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS (N=73) | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA (N=72)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF/VI 100/25 µg QD Via ELLIPTA + Placebo BID Via DISKUS (N=73) | FP 250 µg BID Via DISKUS + Placebo QD Via ELLIPTA (N=72)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT02730351/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02730351/SAP_001.pdf